CLINICAL TRIAL: NCT06822582
Title: A Pelvic Health eModule to Address Urogenital Impairments After Breast and Gynecologic Cancer: a Pilot Prospective Interventional Study
Brief Title: Pelvic Health Rehabilitation After Breast and Gynecologic Cancer
Acronym: GYVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-13-2025-3199
Record Dates: First submitted 2025-01-29; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Gynecologic Cancers; Breast Cancer Female; Incontinence; Incontinence Bowel; Sexual Dysfunction; Vaginal Atrophy, Sexual Dysfunction, Vaginal Dryness, Dyspareunia; Constipation
Keywords: pelvic health; telerehabilitation; supportive cancer care
MeSH Terms: conditions — Encopresis; Sexual Dysfunction, Physiological; Dyspareunia; Constipation

STUDY DESIGN:
Intervention Model Description: Pilot interventional prospective cohort design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pelvic Health Module (Experimental): Participants from the experimental (single) arm will partake in a 12-week intervention involving weekly live online group exercises and educational sessions in French or English. The sessions will be led and supervised by a registered physiotherapist with expertise in pelvic health.
  Interventions: Behavioral: Pelvic Health Module

INTERVENTIONS:
Behavioral: Pelvic Health Module — Telerehabilitation program involving pelvic floor exercises, education and counselling.

SUMMARY:
The GYVE study aims at testing an online program (eModule) to help people who have had breast or gynecologic cancer and are experiencing pelvic health issues like urinary incontinence and pain during sex. These cancers and their treatments can cause significant pelvic health problems, affecting daily life and quality of life. Physiotherapy can help, but access is often limited due to costs and other barriers. The study will involve 20 participants from Quebec and Edmonton, who will take part in a 12-week program with weekly online group sessions led by a physiotherapist. Topics include pelvic floor muscle training, use of vaginal moisturizers, hydration, diet, and pain management. Led by experts in cancer rehabilitation and pelvic health, the study aims to provide valuable information on the feasibility and effectiveness of the eModule, potentially leading to broader implementation to help more people with lived experience of cancer.

DETAILED DESCRIPTION:
The GYVE study aims at testing a new online program (eModule) designed to help people who have had breast or gynecologic cancer and are experiencing pelvic health issues such as urinary incontinence and pain during sex. These cancers are common and can cause pelvic health problems due to treatments like surgery, radiation, and hormone therapy. Many people treated for these cancers experience issues that affect their daily lives and quality of life. Physiotherapy for pelvic health can help, but access to these services is often limited due to costs, travel, and other barriers. The study's goals are to see if the new eModule is practical and well-received by participants and to check if it helps reduce pelvic health problems. More specifically, this study aims to:

Obj 1) Evaluate the feasibility and the acceptability of implementing the new eModule, as perceived by people treated for breast or gynecological cancer.

Obj 2) Explore the preliminary effectiveness of the new eModule in reducing urogenital impairments.

The hypothesis is that the eModule will be practical and well-liked, with at least 70% of participants completing the study and over 85% reporting high satisfaction. The study will be conducted in Quebec and Edmonton with 20 participants who have had breast or gynecologic cancer and are experiencing pelvic health issues. The eModule will last 12 weeks and include weekly online group sessions led by a physiotherapist, covering topics like pelvic floor muscle training, use of vaginal moisturizers, hydration, diet, and pain management. Participants will complete questionnaires before, during, and after the program to measure its impact. Outcomes measured will include feasibility (session attendance and study completion), acceptability (participant satisfaction), and effectiveness (changes in pelvic health issues). The study will follow ethical guidelines to protect participants' privacy and ensure their informed consent.

The study is led by experts in cancer rehabilitation and pelvic health from various Canadian institutions and will take place over several months, with phases for preparation, recruitment, intervention, data collection, and analysis. If successful, this study will provide valuable information on the feasibility and effectiveness of the eModule, potentially leading to larger studies and broader implementation to help more people with lived experience of cancer.

ELIGIBILITY:
Inclusion Criteria:

* be >18 years of age;
* have received a diagnosis of breast or gynecological (endometrial, cervical, ovarian, vulvar or vaginal) cancer (Stage I-IV) ;
* be on active cancer treatment or have completed any cancer treatment (surgery and/or radiation therapy and/or chemotherapy) within the last 3 years;
* be able to provide informed written consent in English or French;
* have a urogenital dysfunction, as screened by a score of ≥ 2 on the Pelvic Floor Bother Questionnaire.

Exclusion Criteria:

* do not have regular access to internet, to a smart device or a computer, at home.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Perceived effectiveness of the intervention | From enrollment to the end of intervention at 12 weeks
  The Patient Global Impression of Change scale will be used to determine the extent to which the intervention is perceived as likely to remedy urogenital deficiencies.

OTHER OUTCOMES:
Adherence Rate | From enrollment to the end of intervention at 12 weeks
  number of intervention sessions attended/participant
Attrition rate | From enrollment to the end of intervention at 12 weeks
  number of participants who did not complete participation / those who did.
International Consultation on Incontinence Questionnaire | From enrollment to the end of intervention at 12 weeks
  a modular questionnaire for urinary symptoms (12 items) and bowel symptoms (20 items).
Vulvar Pain Assessment Questionnaire | From enrollment to the end of intervention at 12 weeks
  a 38-item questionnaire to assess vulvar pain intensity
Female Sexual Function Index | From enrollment to the end of intervention at 12 weeks
  a 19-item multidimensional questionnaire to assess six domains of sexual functioning: desire, arousal, lubrication, orgasm, satisfaction, and pain.
Perceived Self-Efficacy scale | From enrollment to the end of intervention at 12 weeks
  modified from the self-efficacy for chronic disease management questionnaire, a 6-item survey to determine a person's perceived overall ability to cope with symptoms in various challenging or stressful situations.
Program's acceptability | From enrollment to the end of intervention at 12 weeks
  questions developed in connection with program acceptability (Relevance of content, Perceived burden, Appropriateness of intervention and sense of safety, Usability, Geographical accessibility, Satisfaction with ease of access to intervention, Previous access to services, Barriers, and Perceived best time in cancer care trajectory)

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - Centre interdisciplinaire de recherche en réadaptation et intégration sociale, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Undecided